CLINICAL TRIAL: NCT07366866
Title: A Single-center, Randomized, Double-blind, Placebo-controlled, Dose-escalation Phase 1 Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of a Single Subcutaneous Injection of GenSci136 for Injection in Healthy Adult Participants in China.
Brief Title: A Study of Safety, Tolerability, PK, and PD of Subcutaneous GenSci136 in Healthy Adults.
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Changchun GeneScience Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: GenSci136-101
Record Dates: First submitted 2026-01-07; First posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Autoimmune Disease
MeSH Terms: conditions — Autoimmune Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GenSci136 (Experimental): Single ascending doses of GenSci136 administered subcutaneously (SC).
  Interventions: Drug: GenSci136
- Placebo (Placebo Comparator): Administered SC.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GenSci136 — Administered SC.
  Arms: GenSci136
Drug: Placebo — Administered SC.
  Arms: Placebo

SUMMARY:
This study is designed to evaluate the safety, tolerability, PK and PD of GenSci136 in a randomized, double-blind, placebo-controlled trial involving healthy adult participants.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, aged 18 to 45 years (both inclusive) at the time of signing informed consent form (ICF).
2. Male body weight ≥ 50 kg or female body weight ≥ 45 kg; BMI between 18-28 kg/m2 (both inclusive) at screening.
3. Males of reproductive age and females of childbearing potential must agree to take highly effective contraceptive methods from screening to the end of the study, and have no plans for conception, sperm donation, or egg donation; females of childbearing potential must have a negative pregnancy test at screening/baseline period and are not breastfeeding.
4. Able to understand the trial procedures, voluntarily participate in the trial, understand and voluntarily sign the ICF, be able to follow all the trial requirements and complete the study.

Exclusion Criteria:

1. Known hypersensitivity to GenSci136 or any of the excipients contained in the GenSci136 formulation, or history of serious hypersensitivity reactions to any drug, compound, food, or other substance, or an allergic constitution.
2. Presence of tattoo, sunburn, scar or any other factors that may interfere with the assessment of the injection site at the intended injection area.
3. A history or presence of other significant metabolic, dermatologic, hepatic, renal, hematologic, cardiovascular, gastrointestinal, psychoneurological, respiratory, and/or other major disease that, in the opinion of the investigator, would affect the evaluation of the study.
4. Any major surgery within 3 months before screening, plan to undergo elective surgery during the study period, or have a history of any surgery that may affect the absorption, distribution, metabolism or excretion of the IMP.
5. Positive result of alcohol breath test, or drug abuser, or use of soft drugs (such as marijuana) within 3 months prior to screening, or use of hard drugs (such as cocaine and ketamine) within 1 year prior to screening, or positive for drug screening [including but not limited to morphine, ketamine, dimethyldioxyamphetamine, methamphetamine, tetrahydrocannabinol, and cocaine].
6. Participants judged by the investigator to be ineligible for other reasons.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2026-04-28 (Estimated); Primary Completion 2027-02-07 (Estimated); Study Completion 2027-03-09 (Estimated)

PRIMARY OUTCOMES:
● Incidence and severity of treatment-emergent adverse events (TEAEs) ● Incidence and severity of serious adverse events (SAEs) | Day1-Day113

SECONDARY OUTCOMES:
Serum Concentration of free GenSci136/total GenSci136 | Day1-Day113
  Serum concentrations at different time points will be listed and summarized by descriptive statistics.
Maximum serum concentration (Cmax) | Day1-Day113
  PK parameters will be analyzed by non-compartmental analysis with WinNonlin@ version 8.3 or above.
Time to maximum serum concentration (Tmax) | Day1-Day113
  PK parameters will be analyzed by non-compartmental analysis with WinNonlin@ version 8.3 or above.
Area under the concentration-time curve from the time zero to last measurable concentration (AUC0-t) | Day1-Day113
  PK parameters will be analyzed by non-compartmental analysis with WinNonlin@ version 8.3 or above.
Area under concentration-time from time zero to infinity (AUC0-inf) | Day1-Day113
  PK parameters will be analyzed by non-compartmental analysis with WinNonlin@ version 8.3 or above.
Terminal elimination half-life (t1/2) | Day1-Day113
  PK parameters will be analyzed by non-compartmental analysis with WinNonlin@ version 8.3 or above.
Clearance (CL/F) | Day1-Day113
  PK parameters will be analyzed by non-compartmental analysis with WinNonlin@ version 8.3 or above.
Apparent volume of distribution (Vd/F) | Day1-Day113
  PK parameters will be analyzed by non-compartmental analysis with WinNonlin@ version 8.3 or above.
● Changes from baseline in free and total a proliferation inducing ligand (APRIL) levels; ● Changes from baseline in free and total B-cell activating factor (BAFF) levels. | Day1-Day113
Incidence and the time of anti-drug antibody (ADA) positive after GenSci136 administration. | Day1-Day113

CONTACTS AND LOCATIONS:
Locations (1):
- Huashan Hospital, Shanghai, Shanghai Municipality, China